CLINICAL TRIAL: NCT05452083
Title: Postoperative External Beam Whole Breast or Chest Wall Irradiation of Patients With Breast Cancer in Extreme Hypofractionation.
Brief Title: Postoperative Radiation of Patients With Breast Cancer in Extreme Hypofractionation.
Status: Not yet recruiting | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Claudia Schweizer, Dr. med. Claudia Schweizer, University of Erlangen-Nürnberg Medical School
Other Study IDs: ExtremeHypofractionationBreast
Record Dates: First submitted 2022-04-22; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood withdrawals for dynamic immune status
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of treatment toxicity of extreme hypofractionation of the whole breast in five fractions of 5.2 Gy in five consecutive workdays.

DETAILED DESCRIPTION:
The focus of this phase 2-trial is set on feasibility as well as early and late toxicity rates. One possible disadvantage of extreme hypofractionation could be an increased rate of fibrosis within the irradiated region. Therefore, a closer look will be taken with this prospective trial.

In addition, we are planning an accompanying translational research program since hypofractionated schedules are suggested to be more immunogenic in breast cancer.

Secondary objectives therefore are: cosmetic outcome, local tumor control, quality of life, dynamic immune status, importance of tumor infiltrating immune cells, overall survival, disease-free survival, feasibility of breath-hold radiation technique.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast cancer or ductal carcinoma in situ (DCIS)
* pT-category pT0-3
* complete resection (R0)
* Absence of distant metastasis (M0)
* Absence of contralateral breast cancer/ DCIS
* Karnofsky Performance Score ≥ 60%
* Age ≥ 18 years at time of study entry
* Written informed consent

Exclusion Criteria:

* All patients not fulfilling inclusion criteria
* Morbus Paget or pathological skin infiltration
* Earlier or synchronous breast cancer
* Pregnant or breast-feeding women
* Increased radiosensitivity or any genetic disposition for increased radiosensitivity, e.g. ataxia telangiectatica
* Judgement by the investigator that the patient is unlikely to comply with study procedures and requirements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with breast cancer after complete resection and the indication for postoperative radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2035-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and grade of Treatment related adverse events according to the Common Terminology Criteria for Adverse Events (CTCAE 5.0) | 08/2022 - 07/2035
  Evaluation during treatment and at each follow-up visit up to 10 years

SECONDARY OUTCOMES:
Cosmetic results according to the Harvard-scale | 05/2022 - 04/2035
  Clinical evaluation of the irradiated breast at each follow-up up to 10 years according to the Harvard-scale (patient's and physician's view)
In-breast recurrence rate | 05/2022 - 04/2035
  Evaluation at each follow-up up to 10 years via regular examinations including mammography/ ultrasound
Quality of life during and after treatment using the patient-reported questionnaires EORTC QLQ-C30 and QLQ-BR23 | 05/2022 - 04/2035
  Evaluation of patient's quality of life from inclusion to each follow-up up to 10 years via standardized questionnaires: European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire QLQ-C30 and the breast-orientated QLQ-BR23
Immune status analysis: Immunophenotyping using peripheral blood at several time points | 05/2022 - 04/2027
  Withdrawals of whole blood (plasma and serum) before the first irradiation until one year after the treatment. Immunophenotyping by a modular multicolor flow cytometry-based method. Furthermore, whole exome sequencing/RNASeq on already obtained tissue from the breast surgery.
Overall survival | 05/2022 - 04/2035
  Evaluation at each follow-up up to 10 years
Evaluation of feasibility of breath-hold radiation technique throughout the treatment time | 05/2022 - 04/2025
  Evaluation of patient's capability to follow breathing commandos during planning-CT scan and each application of radiotherapy